CLINICAL TRIAL: NCT05385952
Title: A Prospective, Multicenter, Randomized Clinical Investigation Evaluating the Safety and Efficacy of GATT-Patch Versus TachoSil for Hemostasis During Open Liver Surgery
Brief Title: GATT-Patch Versus TachoSil in Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GATT Technologies BV (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHF-01-SFT-194
Record Dates: First submitted 2022-04-29; First posted 2022-05-23 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Intraoperative Bleeding; Hemorrhage, Surgical; Liver Diseases
Keywords: Hemostatic patch; GATT-Patch; TachoSil; Liver surgery; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Liver Diseases | interventions — TachoSil

STUDY DESIGN:
Intervention Model Description: Randomization 2:1
Who Masked: Participant
Masking Description: Patients will be blinded to randomized treatment and treatment used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- GATT-Patch (currently named ETHIZIA) (Experimental): Hemostatic patch
  Interventions: Device: GATT-Patch (currently named ETHIZIA)
- TachoSil (Active Comparator): Hemostatic patch
  Interventions: Drug: TachoSil

INTERVENTIONS:
Device: GATT-Patch (currently named ETHIZIA) — GATT-Patch (currently named ETHIZIA) is a sterile, flexible and resorbable hemostatic sealing patch. It presents as a blue, soft, flexible, porcine gelatin fiber-based carrier impregnated with an NHS-POx / NU-POx granulate. GATT-Patch measures 10 cm long by 5 cm wide. GATT-Patch is active and can be applied on both sides. Blue color is an aid to visualize GATT-Patch when applied onto a bleeding location.
  GATT-Patch is indicated for use as an adjunct to hemostasis in surgery for minimal, mild or moderate bleeding sites when control of bleeding by standard surgical techniques (such as suture, ligature or cautery) is ineffective or impractical. GATT-Patch is intended to be used for management of hemorrhage during surgeries on the liver.
  Arms: GATT-Patch (currently named ETHIZIA)
Drug: TachoSil — TachoSil is a topical fibrin sealant patch consisting of human fibrinogen and human thrombin coated onto an equine collagen sponge.
  TachoSil is a fibrin sealant patch indicated for use with manual compression in adult and pediatric patients as an adjunct to hemostasis in cardiovascular and hepatic surgery, when control of bleeding by standard surgical techniques (such as suture, ligature or cautery) is ineffective or impractical.
  Arms: TachoSil

SUMMARY:
This is a pre-market, prospective, randomized (2:1), multicenter, multi-national pivotal clinical investigation. The purpose of this investigation is to determine the clinical safety and performance of GATT-Patch as compared with TachoSil for the management of minimal, mild, or moderate bleeding during elective open liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo elective open surgery on the liver;
* Subject is willing and able to give written informed consent for the clinical investigation participation;
* Subjects is 22 years of age or older at the time of enrollment; and
* Subject has been informed of the nature of the clinical investigation.

A subject must meet all of the following intra-operative inclusion criteria to be enrolled into the clinical investigation:

* Subject in whom the Investigator is able to identify a target bleeding site at the liver resection plane for which any applicable conventional means for hemostasis (e.g. suture, ligature or cautery) are ineffective or impractical, and the choice is made to use a hemostatic agent to stop the bleeding; and
* Subject has a target bleeding site with a SBSS of 1, 2, or 3 (e.g. reflecting minimal, mild or moderate bleeding severities).

Exclusion Criteria:

* The target bleeding site is from a large defect in an artery or vein that requires vascular reconstruction with maintenance of vessel patency;
* Subject is scheduled to undergo surgery on other organs than the liver and its associated biliary and vascular system; • Subject is scheduled to undergo a staged liver surgery procedure (e.g., Associating Liver Partition and Portal vein ligation for Staged hepatectomy [ALPPS])
* Subject is taking multiple antithrombotic therapies in therapeutic dosage up to the time of surgery, but allowing exclusive use of acetylsalicylic acid;
* Subject has platelet count <100 x 109/L, an activated partial thrombin time of >100s, or international normalized ratio >2.5;
* Subject has a total bilirubin level of ≥2.5 mg/dl;
* Subject is pregnant, planning on becoming pregnant or actively breastfeeding during the 3-month follow-up period;
* Subject has a known hypersensitivity to brilliant blue (FD&C Blue #1), porcine gelatin, or horse proteins;
* Subject who has religious objections to receiving products with components of animal (porcine or equine) or human origin;
* Subject has an active or suspected infection at the bleeding site;
* Subject in whom the investigational device will be used at the site of a synthetic graft or patch implant;
* Subject has a life expectancy of less than 3 months;
* Subject has a documented severe congenital or acquired immunodeficiency;
* Subject has had or has planned to receive any organ transplantation;
* Subject undergoes surgery with the indication of being a living liver donor;
* Subject is currently participating or has participated in another clinical investigation within the past 30 days that may affect the endpoints of the study, such as trials related to the surgical procedure, and on anti-coagulation;
* Subject is not appropriate for inclusion in the clinical investigation, per the medical opinion of the Investigator; and
* Subject has any incidental (pre- and peri-operative) findings deemed by the Investigator to potentially jeopardize the safety or welfare of the subject.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Rate of hemostasis at 3 minutes without rebleeding at the 10-minute time point | During surgical procedure
  SBSS 0

SECONDARY OUTCOMES:
Mean time to hemostasis (seconds) | During surgical procedure
  SBSS 0
Kaplan-Meier estimated distribution of time to hemostasis | During surgical procedure
  SBSS 0
Rate of subjects with treatment failure | During surgical procedure
  SBSS 1-5 at the 10 minute timepoint
Rate of subjects with rebleeding after 10 minutes but before subject closure | During surgical procedure
  SBSS 1-5 after initially SBSS 0
Rate of subjects with hemostasis at 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 360, 420, 540 and 600 seconds | During surgical procedure
  SBSS 0-5

OTHER OUTCOMES:
Procedure duration | During surgical procedure
  Time in minutes
Estimated blood loss | During surgical procedure
  mL
Number and type of blood transfusions | During surgical procedure
  Platelets, Erythrocytes, Plasma
Number and type of blood transfusions | During hospitalization up to hospital discharge after the surgical procedure, estimated up to 30 days
  Platelets, Erythrocytes, Plasma
Mean duration of ICU stay | From surgery to discharge from the ICU, estimated up to 30 days
  Time in hours
Mean total hospitalization time | During hospitalization up to hospital discharge after the surgical procedure, estimated up to 30 days
  Time in days
Aspect of postoperative drainage | During hospitalization up to hospital discharge after the surgical procedure, estimated up to 30 days
  Serous, sanguineous, serosanguineous, other Sanguineous Serosanguinous Serous, Sanguineous, Serosanguineous, Purulent, Other
Rate of subjects requiring reoperation | During postoperative 3-months follow-up
  Occurrence yes/no
Rate of subjects with liver resection surface complications on ultrasound | At 6 weeks follow-up visit
  Fluid collection, biloma, hematoma, patch encapsulation, patch rolling up on the surface
Amount of hemostatic material needed versus bleeding surface | During surgical procedure
  cm2 patch per cm2 bleeding
System Usability Score (SUS) user satisfaction questionnaire | At completion of the surgical procedure, at day 0
  Likert scale (strongly disagree, disagree, neutral, agree, strongly agree) with (strongly) agreeing meaning a better outcome for uneven questions and (strongly) disagreeing meaning a better outcome for even questions
GATT-Patch device-specific user satisfaction questionnaire | At completion of the surgical procedure, at day 0
  Likert scale (strongly disagree, disagree, neutral, agree, strongly agree) with (strongly) agreeing meaning a better outcome
Local recurrence of liver cancer at the resection | 5 years
  Occurrence yes/no
Cancer-free survival | 5 years
  Occurrence yes/no
Overall survival | 5 years
  Occurrence yes/no

CONTACTS AND LOCATIONS:
Overall Officials: James Guarrera, Principal Investigator — Rutgers New Jersey Medical School, Newark, NJ, USA; Hans de Wilt, Principal Investigator — Radboud University Medical Center
Locations (10):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Washington University, St Louis, Missouri
  - Rutgers University, Newark, New Jersey
  - Weill-Cornell, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Intermountain Healthcare, Murray, Utah
- Heidelberg University Hospital, Heidelberg, Germany
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boerman MA, Roozen E, Sanchez-Fernandez MJ, Keereweer AR, Felix Lanao RP, Bender JCME, Hoogenboom R, Leeuwenburgh SC, Jansen JA, Van Goor H, Van Hest JCM. Next Generation Hemostatic Materials Based on NHS-Ester Functionalized Poly(2-oxazoline)s. Biomacromolecules. 2017 Aug 14;18(8):2529-2538. doi: 10.1021/acs.biomac.7b00683. Epub 2017 Jul 25. PMID 28699748
- [Background] Roozen EA, Warle MC, Lomme RMLM, Felix Lanao RP, van Goor H. New polyoxazoline loaded patches for hemostasis in experimental liver resection. J Biomed Mater Res B Appl Biomater. 2022 Mar;110(3):597-605. doi: 10.1002/jbm.b.34938. Epub 2021 Sep 18. PMID 34536065